CLINICAL TRIAL: NCT02798003
Title: Analysis of Food Reward System in Cachexia Induced by Acute or Chronic Disease
Brief Title: Food Reward in Cachexia Induced by Acute or Chronic Disease
Status: Terminated | Type: Observational
Why Stopped: Not feasible to include the needed patients
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NL54799.068.15
Record Dates: First submitted 2016-03-31; First posted 2016-06-14 (Estimated); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Cachexia; Chronic Obstructive Pulmonary Disease; Non-small Cell Lung Cancer; Pancreatic Cancer
Keywords: Cachexia; Food reward
MeSH Terms: conditions — Cachexia; Pulmonary Disease, Chronic Obstructive; Carcinoma, Non-Small-Cell Lung; Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Cachectic cancer patients: Cachectic cancer patients, including non-small cell lung cancer (NSCLC) and gastro-intestinal cancer. The study participants will undergo fMRI scanning.
  Interventions: Other: Functional magnetic resonance imaging (fMRI)
- Non-cachectic cancer patients: Non-cachectic cancer patients, including NSCLC and gastro-intestinal cancer. The study participants will undergo Functional magnetic resonance imaging (fMRI) scanning.
  Interventions: Other: Functional magnetic resonance imaging (fMRI)
- Cachectic COPD patients: Diagnosis of Chronic Obstructive Pulmonary Disease (COPD) consistent with the Global Initiative for Chronic Obstructive Lung Disease (GOLD) criteria. The study participants will undergo fMRI scanning.
  Interventions: Other: Functional magnetic resonance imaging (fMRI)
- Non-cachectic COPD patients: Diagnosis of COPD consistent with the Global Initiative for Chronic Obstructive Lung Disease (GOLD) criteria. The study participants will undergo fMRI scanning.
  Interventions: Other: Functional magnetic resonance imaging (fMRI)

INTERVENTIONS:
Other: Functional magnetic resonance imaging (fMRI) — The food-cue elicited response in the reward-circuitry of the brain will be assessed by using fMRI. This technique is based on different magnetic properties of oxygenated and deoxygenated blood. Increased neuronal activity causes an increase in blood flow. Thereby, neuronal activity is indirectly reflected by changes in blood oxygenation level-dependent (BOLD) contrast.

SUMMARY:
To study activity in the reward-circuitry of the brain in patients suffering from cachexia induced by cancer or chronic disease.

DETAILED DESCRIPTION:
The activity in the food reward-circuitry of the brain in patients suffering from cachexia induced by cancer (lung cancer or pancreatic cancer) or chronic disease (chronic obstructive pulmonary disease) will be analysed by using functional magnetic resonance imaging. In addition, the role of the peripheral satiety hormones will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* For cachectic patients: weight loss exceeds 5% of total body weight over the past 6 months, or >2% when body mass index is <20 kg/m2
* For non-cachectic patients: no weight loss of ≥5% during the last 6 months
* Non-small cell lung cancer or gastro-intestinal cancer, pathology proven or diagnosis of COPD consistent with the Global Initiative for Chronic Obstructive Lung Disease (GOLD) criteria

Exclusion Criteria:

* Contra-indications for fMRI examination (operation to your head or brain in the past; implanted electronic devices, for instance a pacemaker, neurostimulator, cochlear or hearing implant; insulin pump under your skin; Pregnant subjects, claustrophobia; pregnancy; metal parts in your body (except from teeth filling and connectors): implants; brain vessel clamps, prostheses, intra-uterine device, metal splinter in the eye, metal braces or other metal objects, permanent eye make-up)
* Psychiatric or other disorders likely to impact on informed consent
* Presence of brain metastasis (screening is not mandatory)
* Medical history of cerebrovascular accident, brain tumour, brain metastasis
* Previous radiotherapy to brain, both stereotactic and whole brain radiotherapy
* Memory problems
* Current use of tube feeding or parental nutrition
* Patients with an active second malignancy
* Patients unable to lie still for 2 hours
* Unable to complete the cognitive task
* Pre-existing swallowing difficulties
* Allergy to gluten-, milk- or wheat products
* Self-reported hyperthyroidism
* Self-reported diabetes mellitus
* Current use of appetite stimulant medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Four groups will be included:
  1. Cachectic cancer patients, including NSCLC and gastro-intestinal cancer
  2. Non-cachectic cancer patients, including NSCLC and gastro-intestinal cancer
  3. Cachectic COPD patients
  4. Non-cachectic COPD patients
  Individuals of all groups will be gender and age matched. In addition, COPD patients will be matched for FEV1.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2022-02-18 (Actual); Study Completion 2022-02-18 (Actual)

PRIMARY OUTCOMES:
Reward-related activity in response to food cues, as indicated by Blood Oxygenation Level Dependent (BOLD) values in specified brain areas related to food reward. | 2 years

SECONDARY OUTCOMES:
Dietary intake assessed by a food diary | 2 years
Blood parameters: glucose (mmol/L) | 2 years
Blood parameters: insulin (pmol/L) | 2 years
Blood parameters: leptin (ug/L) | 2 years
Blood parameters: ghrelin (pg/mL) | 2 years
Blood parameters: glucagon-like peptide-1 (pmol/L) | 2 years

OTHER OUTCOMES:
Anthropometrical characteristics: body mass index (kg/m2) | 2 years
Other relevant co-variables: current medical status (charlson co-morbidity index scale) | 2 years
Other relevant co-variables: World Health Organization performance score (WHO PS) | 2 years
Other relevant co-variables: pulmonary function (Forced Expiration Volume in 1 second [FEV1] in % predicted) | 2 years
Other relevant co-variables: pulmonary function (diffusing capacity of the lungs for carbon monoxide [DLCO] in % predicted) | 2 years
Other relevant co-variables: weight change past 6 months (kg) | 2 years
Other relevant co-variables: self-reported smoking status of all 44 participants (current, former, never, in pack years) | 2 years
Changes in food preferences assessed by the Functional Assessment of Anorexia/Cachexia Therapy (FAACT) | 2 years
Cognitive functioning assessed by Mini-Mental State Examination (MMSE) | 2 years
Cognitive functioning assessed by Cognitive Failure Questionnaire (CFQ) | 2 years
Presence of depression and anxiety assessed by the Hospital Anxiety and Depression Scale (HADS) | 2 years
General wellbeing assessed by the European Organization for Research and Treatment of Cancer (EORTC) c30 questionnaire | 2 years
Inflammatory parameters: c-reactive protein (ml/L) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Annemie Schols, PhD, Principal Investigator — Maastricht UMC
Locations (1):
- Maastricht UMC, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided